CLINICAL TRIAL: NCT02324751
Title: A Phase IIb, Observer-blind, Randomised Controlled Trial to Assess the Immunogenicity and Protective Efficacy of Vi Conjugated (Vi-TCV) and Unconjugated (Vi-PS) Polysaccharide Vaccines in Preventing Typhoid Infection Compared to a Control Vaccine (Meningococcal ACWY), Using a Human Challenge Model of Typhoid Infection
Brief Title: Vaccines Against Salmonella Typhi
Acronym: VAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OVG 2014/08
Record Dates: First submitted 2014-12-02; First posted 2014-12-24 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2018-02

CONDITIONS: Typhoid Fever; Enteric Fever
MeSH Terms: conditions — Typhoid Fever | interventions — Vi polysaccharide vaccine, typhoid; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vi-TCV (Experimental): Single intramuscular injection
  Interventions: Biological: Vi-TCV
- Vi-PS Vaccine (Active Comparator): Single intramuscular injection
  Interventions: Biological: Vi-PS Vaccine
- Control (Men ACWY) (Other): Single intramuscular injection
  Interventions: Biological: Control (Men ACWY)

INTERVENTIONS:
Biological: Vi-TCV — Each 0.5mL vaccine dose contains 25μg of purified Vi capsular polysaccharide (S. Typhi Ty2 strain) conjugated to non-toxic tetanus toxoid. The vaccine will be administered 28 days prior to typhoid challenge
  Other Names: Typbar-TCV
  Arms: Vi-TCV
Biological: Vi-PS Vaccine — Each 0.5 mL vaccine dose contains 25 μg of purified Vi capsular polysaccharide (S. Typhi Ty2 strain). The vaccine will be administered 28 days prior to typhoid challenge
  Other Names: TYPHIM Vi
  Arms: Vi-PS Vaccine
Biological: Control (Men ACWY) — Each vaccine dose contains N. meningitidis oligosaccharides (10μg MenA oligosaccharide, 5μg of each of MenC, Men Y and MenW-135 oligosaccharides) conjugated to 32.7 μg to 64.1μg Diphtheria CRM197 protein with residual formaldehyde dose less than 0.30μg. The vaccine will be administered 28 days prior to typhoid challenge
  Other Names: MENVEO
  Arms: Control (Men ACWY)

SUMMARY:
Using an established model of human typhoid infection, whereby healthy adults are deliberately exposed to typhoid-causing bacteria, the investigators will determine how effective a new typhoid conjugate vaccine (Vi-TCV) is in preventing infection. The new typhoid vaccine will be compared with a control vaccine (meningococcal ACWY). The protective effect of a currently used typhoid polysaccharide vaccine (Vi-PS) will also be studied and compared with the control vaccine using this model of typhoid infection.

A second component of this study will involve vaccinating 15-20 participants with Vi-PS. Serum will be obtained prior to vaccination and 4-6 weeks after vaccination. The post-vaccination serum will be pooled and used to create an anti-Vi IgG serum standard.

DETAILED DESCRIPTION:
Typhoid fever is an infection caused by a bacterium, Salmonella Typhi, that only causes disease in humans. It is transmitted faecal-orally and causes more than 22 million infections every year in developing countries, such as areas of Asia, Africa and South America, where access to clean drinking water and sanitation facilities is limited. Although typhoid fever is treatable with effective antibiotics, there are more than 200,000 deaths every year in these resource-limited regions.

Salmonella Typhi could be eradicated but improving sanitation and living conditions in endemic regions is difficult. Vaccination to prevent the transmission of Salmonella Typhi could significantly reduce the burden of disease. The currently licensed typhoid vaccines are only moderately effective in preventing infection in people who have been immunised and no vaccines are licensed for use in young children. Novel typhoid vaccines have been developed to overcome these problems, but more research and information is needed to study how well these vaccines work before they can be routinely used.

This study proposes to investigate the protective effect of a novel typhoid vaccine (typhoid Vi polysaccharide capsule - tetanus toxoid conjugate vaccine) using a human challenge model of typhoid infection. Healthy adults will be vaccinated with the novel typhoid vaccine, a currently used typhoid vaccine (Vi polysaccharide capsule vaccine) or a control vaccine. One month after vaccination, participants will be exposed to live Salmonella Typhi by drinking a solution containing the bacteria. Participants will then be closely monitored to determine which participants develop infection and which are protected. In addition to assessing the protective effect of conjugated and unconjugated typhoid vaccines, the effect the vaccines have on the immune system and on the clinical course of typhoid infection will also be studied.

It is hoped that the knowledge gained from this study will contribute to the use of vaccines against Salmonella Typhi to help control this preventable disease.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all of the following criteria to be considered eligible for the study:

* Agree to give informed consent for participation in the study.
* Aged between 18 and 60 years inclusive at time of vaccination.
* In good health as determined by medical history, physical examination and clinical judgment of the study team.
* Agree (in the study team's opinion) to comply with all study requirements, including capacity to adhere to good personal hygiene and infection control precautions.
* Agree to allow his or her General Practitioner (and/or Consultant if appropriate), to be notified of participation in the study.
* Agree to allow study staff to contact his or her GP to access the participant's vaccination records.
* Agree to allow Public Health England to be informed of their participation in the study.
* Agree to give his or her close contacts written information informing them of the participant's involvement in the study and offer them voluntary screening for S. Typhi carriage.
* Agree to have 24-hour contact with study staff during the four weeks post challenge and are able to ensure that they are contactable by mobile phone for the duration of the challenge period until antibiotic completion.
* Have internet access to allow completion of the e-diary and real-time safety monitoring.
* Agree to avoid antipyretic/anti-inflammatory treatment from the time of challenge (Day 0) until advised by a study doctor or until 14 days after challenge.
* Agree to provide their National Insurance/Passport number for the purposes of TOPS registration and for payment of reimbursement expenses.

Exclusion Criteria:

The participant will not be enrolled if any of the following apply:

* History of significant organ/system disease that could interfere with trial conduct or completion. Including, for example, but not restricted to: Cardiovascular, respiratory, haematological, endocrine, Renal/bladder, biliary tract, gastro-intestinal, neurological, metabolic, autoimmune or infectious disease. Or Psychiatric illness requiring hospitalisation or known or suspected drug and/or alcohol misuse
* Have any known or suspected impairment of immune function, alteration of immune function, or prior immune exposure that may alter immune function to typhoid infection
* Moderate or severe depression or anxiety as classified by the Hospital Anxiety and Depression Score at screening or challenge that is deemed clinically significant by the study doctors .
* Weight less than 50kg
* Presence of implants or prosthesis.
* Anyone taking long-term medication that may affect symptom reporting or interpretation of the study results.
* Contraindication to ciprofloxacin or macrolide antibiotics.
* Female participants who are pregnant, lactating or who are unwilling to ensure that they or their partner use effective contraception one month prior to challenge and continue to do so until two negative stool samples, a minimum of 2 weeks after completion of antibiotic treatment, have been obtained.
* Occupations involving:

  * Direct contact with young children attending pre-school groups or nursery or aged under 2 years, or
  * Direct contact with highly susceptible patients or persons in whom typhoid infection would have particularly serious consequences (unless willing to avoid work until demonstrated not to be infected with typhoid in accordance with guidance from Public Health England)
* Occupations involving commercial food handling
* Close household contact with:

  * Young children (defined as those attending pre-school groups, nursery or those aged less than 2 years)
  * Immunocompromised individuals
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study period.
* Participants who have participated in another research study involving an investigational product within the 30 days prior to enrolment
* Detection of any abnormal results from screening investigations (at the clinical discretion of the study team).
* Inability to comply with any of the study requirements
* Any other social, psychological or health issues which, in the opinion of the study staff, may

  * Put the participant or their contacts at risk because of participation in the study,
  * Adversely affect the interpretation of the primary endpoint data,
  * Impair the participant's ability to participate in the study.
* Having previously received any typhoid vaccine
* Having been resident in an enteric fever endemic country for 6 months or more.
* Have previously been diagnosed with laboratory-confirmed typhoid or paratyphoid infection or been given a diagnosis compatible with enteric fever.
* Have participated in previous typhoid or paratyphoid challenge studies
* Have received vaccination with tetanus toxoid containing vaccine within the past 12 months.
* Have any history of allergy to vaccine components
* Have a prolonged corrected QT interval (>450 milliseconds) on ECG screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12-02 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Clinically or microbiologically proven typhoid infection | Up to 14 days after typhoid challenge dose administration
  Clinical (fever >38 degrees for more than 12 hours) or microbiologically (blood culture positive) proven typhoid infection following oral challenge with Salmonella Typhi.

SECONDARY OUTCOMES:
Clinical manifestations of typhoid infection after typhoid challenge as determined by physical examination, participant symptom reporting and microbiological assays | Clinical signs and solicited symptoms occurring during the 21 day period after challenge; microbiological assays and unsolicited symptoms followed up over the course of one year
  In particular comparing control and typhoid vaccination groups regarding time to onset of symptoms, duration of illness, symptom severity, time to onset of bacteraemia, time to onset of stool shedding, and inflammatory response after typhoid challenge
Host immune responses (including Geometric Mean Titres of Salmonella Typhi antigen specific antibodies, antigen specific cell frequencies) at baseline, post-vaccination and post-typhoid challenge time points | From baseline (pre-vaccination) to final follow up visit at one year
Laboratory and high-throughput assays to measure gene expression and protein translation at baseline, post-vaccination and post-challenge time points | From baseline (pre-vaccination) to 28 days after challenge (total duration 2 months)
  To assess variation in genomic response to vaccination with Vi-TCV, Vi-PS and control vaccine and subsequent Salmonella Typhi challenge
Exploratory analysis of blood and faeces samples to investigate novel diagnostic methods for detecting Salmonella Typhi infection | From time of challenge until time of typhoid diagnosis (maximum time frame of 14 days)
Assessment of the number of participants reporting solicited local and systemic reactions, and unsolicited adverse events following vaccination with Vi-TCV | From time of vaccination until 7 days post-vaccination

OTHER OUTCOMES:
Producing an anti-Vi IgG serum standard from volunteers vaccinated with Vi-PS (Vi polysaccharide vaccine) | From time of vaccination until 4-6 weeks post-vaccination
  Sera obtained at baseline and 4-6 weeks post-vaccination, followed by pooling of post-vaccination sera to form an anti-Vi IgG serum standard

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, FRCPCH, PhD, Principal Investigator — Oxford Vaccine Group, The University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Zhu H, Chelysheva I, Cross DL, Blackwell L, Jin C, Gibani MM, Jones E, Hill J, Truck J, Kelly DF, Blohmke CJ, Pollard AJ, O'Connor D. Molecular correlates of vaccine-induced protection against typhoid fever. J Clin Invest. 2023 Aug 15;133(16):e169676. doi: 10.1172/JCI169676. PMID 37402153
- [Derived] Li K, Dodds M, Spreng RL, Abraha M, Huntwork RHC, Dahora LC, Nyanhete T, Dutta S, Wille-Reece U, Jongert E, Ewer KJ, Hill AVS, Jin C, Hill J, Pollard AJ, Munir Alam S, Tomaras GD, Dennison SM. A tool for evaluating heterogeneity in avidity of polyclonal antibodies. Front Immunol. 2023 Feb 16;14:1049673. doi: 10.3389/fimmu.2023.1049673. eCollection 2023. PMID 36875126
- [Derived] Jin C, Gibani MM, Pennington SH, Liu X, Ardrey A, Aljayyoussi G, Moore M, Angus B, Parry CM, Biagini GA, Feasey NA, Pollard AJ. Treatment responses to Azithromycin and Ciprofloxacin in uncomplicated Salmonella Typhi infection: A comparison of Clinical and Microbiological Data from a Controlled Human Infection Model. PLoS Negl Trop Dis. 2019 Dec 26;13(12):e0007955. doi: 10.1371/journal.pntd.0007955. eCollection 2019 Dec. PMID 31877141
- [Derived] Jin C, Gibani MM, Moore M, Juel HB, Jones E, Meiring J, Harris V, Gardner J, Nebykova A, Kerridge SA, Hill J, Thomaides-Brears H, Blohmke CJ, Yu LM, Angus B, Pollard AJ. Efficacy and immunogenicity of a Vi-tetanus toxoid conjugate vaccine in the prevention of typhoid fever using a controlled human infection model of Salmonella Typhi: a randomised controlled, phase 2b trial. Lancet. 2017 Dec 2;390(10111):2472-2480. doi: 10.1016/S0140-6736(17)32149-9. Epub 2017 Sep 28. PMID 28965718
- See also: Related Info — https://journals.plos.org/plosntds/article?id=10.1371/journal.pntd.0007955
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8304662/